CLINICAL TRIAL: NCT01245348
Title: Relative Effectiveness of Schizophrenia Therapy (REST) Study
Brief Title: Relative Effectiveness of Schizophrenia Therapy Study
Acronym: REST
Status: Completed | Type: Observational
Sponsor: Medco Health Solutions, Inc. (Industry)
Collaborators: SureGene, LLC (Industry)
Responsible Party: Principal Investigator, Kelly Parsons, Senior Research Manager, Medco Health Solutions, Inc.
Other Study IDs: REST
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; Bipolar Disorder; atypical antipsychotic; adherence; cost effectiveness; pharmacogenetics; mental illness; SULT4A1
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Mental Disorders

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — One milliliter of saliva will be self collected by study subjects for genetic testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Schizophrenia: Patient with schizophrenia
  Interventions: Genetic: SULT4A1-1 genetic test
- Bipolar: Patient with bipolar disorder
  Interventions: Genetic: SULT4A1-1 genetic test

INTERVENTIONS:
Genetic: SULT4A1-1 genetic test — SULT4A1-1 haplotype result (+/-)

SUMMARY:
The purpose of this study is to validate that SULT4A1-1 status stratification improves responses to atypical antipsychotics in schizophrenia and to extend these findings into bipolar disorder.

DETAILED DESCRIPTION:
The total economic burden for schizophrenia (SZ) in the U.S. is estimated to be more than $60 billion annually. A large contributor to the economic burden of this and other chronic mental disorders, including bipolar disorder (BPD), is the exacerbation of symptoms and disability due to lack of drug efficacy. For these disorders, clinicians typically choose a first line antipsychotic therapy without the support of a diagnostic tool; often, patients are switched to another drug after less than six months of treatment due to what is perceived by patients and clinicians as both insufficient efficacy and unacceptable side effects.

Originally, the sulfotransferase family 4A, member 1 (SULT4A1) gene was selected as a biomarker of interest in SZ based on results showing associations between the gene and disease severity. Later on, SULT4A1 gene status was also associated with better efficacy of atypical antipsychotic (e.g. Zyprexa® (olanzapine) and Risperdal® (risperidone)), with respect to both time to discontinuation and quantitative measures of clinical improvement.

In this prospectively designed, non-randomized retrospective study, we will recruit and genotype subjects with schizophrenia or bipolar disorder that were/are new to therapy for any of the four drugs under evaluation. By looking at retrospective and prospective longitudinal medical and pharmacy data stored within the integrated claims database, we will validate the association of the SULT4A1 gene to the efficacy of selected atypical antipsychotic therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age
* Subjects with either a confirmed diagnosis of schizophrenia or bipolar disorder or subjects with self reported schizophrenia or bipolar disorder
* Subjects who were/are new to therapy for olanzapine, risperidone, quetiapine or ziprasidone
* Subjects who are willing and able to provide informed consent

Exclusion Criteria:

* Subjects initially prescribed less than the generally accepted minimally effective dose of the drugs under study
* Subjects with Major Depressive Disorder (MDD) or another psychotic disorder other than schizophrenia or bipolar disorder
* Subjects with catatonic schizophrenia
* Subjects with moderate to severe mental retardation
* Subjects that refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18y/o) with either a schizophrenia or bipolar disorder diagnosis and were/are new to therapy for olanzapine, risperidone, quetiapine or ziprasidone.
Sampling Method: Non-Probability Sample
Enrollment: 1110 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Assess differences in time to discontinuation (TTD) of olanzapine and risperidone therapy between schizophrenia and bipolar disorder subjects (independently) who are SULT4A1-1 haplotype-positive and who are SULT4A1-1 haplotype-negative | 1 year

SECONDARY OUTCOMES:
Assess differences in time to discontinuation (TTD) of quetiapine and ziprasidone therapy between schizophrenia and bipolar disorder subjects (independently) who are SULT4A1-1 haplotype-positive and who are SULT4A1-1 haplotype-negative | 1 year
For each drug under study assess hospitalization rates for psychiatric illness between schizophrenia and bipolar disorder subjects (independently) who are SULT4A1-1 haplotype-positive and who are SULT4A1-1 haplotype-negative | 1 year
Evaluate whether there are differences in time to discontinuation (TTD) of each drug under study between schizophrenia and bipolar disorder subjects (combined) who are SULT4A1-1 haplotype-positive and who are SULT4A1-1 haplotype-negative | 1 year
Evaluate whether there are differences in overall medical spending between schizophrenia and bipolar disorder subjects (independently and combined) who are SULT4A1-1 haplotype-positive and who are SULT4A1-1 haplotype-negative for each drug under study | 1 year
Evaluate whether there are differences in adherence to each drug under study between schizophrenia and bipolar disorder subjects (independently and combined) who are SULT4A1-1 haplotype-positive and who are SULT4A1-1 haplotype-negative | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Parsons, Ph.D., Principal Investigator — Medco Health Solutions, Inc.
Locations (1):
- Medco Health Solutions, Inc., Franklin Lakes, New Jersey, United States

REFERENCES:
- [Background] Nasrallah HA. The case for long-acting antipsychotic agents in the post-CATIE era. Acta Psychiatr Scand. 2007 Apr;115(4):260-7. doi: 10.1111/j.1600-0447.2006.00982.x. PMID 17355516
- [Background] Stroup TS, McEvoy JP, Swartz MS, Byerly MJ, Glick ID, Canive JM, McGee MF, Simpson GM, Stevens MC, Lieberman JA. The National Institute of Mental Health Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) project: schizophrenia trial design and protocol development. Schizophr Bull. 2003;29(1):15-31. doi: 10.1093/oxfordjournals.schbul.a006986. PMID 12908658
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203
- [Background] Sullivan PF, Lin D, Tzeng JY, van den Oord E, Perkins D, Stroup TS, Wagner M, Lee S, Wright FA, Zou F, Liu W, Downing AM, Lieberman J, Close SL. Genomewide association for schizophrenia in the CATIE study: results of stage 1. Mol Psychiatry. 2008 Jun;13(6):570-84. doi: 10.1038/mp.2008.25. Epub 2008 Mar 18. PMID 18347602
- [Background] Liyou NE, Buller KM, Tresillian MJ, Elvin CM, Scott HL, Dodd PR, Tannenberg AE, McManus ME. Localization of a brain sulfotransferase, SULT4A1, in the human and rat brain: an immunohistochemical study. J Histochem Cytochem. 2003 Dec;51(12):1655-64. doi: 10.1177/002215540305101209. PMID 14623933
- [Background] Minchin RF, Lewis A, Mitchell D, Kadlubar FF, McManus ME. Sulfotransferase 4A1. Int J Biochem Cell Biol. 2008;40(12):2686-91. doi: 10.1016/j.biocel.2007.11.010. Epub 2007 Dec 3. PMID 18248844
- [Background] Hildebrandt MA, Carrington DP, Thomae BA, Eckloff BW, Schaid DJ, Yee VC, Weinshilboum RM, Wieben ED. Genetic diversity and function in the human cytosolic sulfotransferases. Pharmacogenomics J. 2007 Apr;7(2):133-43. doi: 10.1038/sj.tpj.6500404. Epub 2006 Jun 27. PMID 16801938
- [Background] Lewis AG, Minchin RF. Lack of exonic sulfotransferase 4A1 mutations in controls and schizophrenia cases. Psychiatr Genet. 2009 Feb;19(1):53-5. doi: 10.1097/YPG.0b013e3283118776. PMID 19125109
- [Background] Brennan MD, Condra J. Transmission disequilibrium suggests a role for the sulfotransferase-4A1 gene in schizophrenia. Am J Med Genet B Neuropsychiatr Genet. 2005 Nov 5;139B(1):69-72. doi: 10.1002/ajmg.b.30222. PMID 16152568
- [Background] Condra JA, Neibergs H, Wei W, Brennan MD. Evidence for two schizophrenia susceptibility genes on chromosome 22q13. Psychiatr Genet. 2007 Oct;17(5):292-8. doi: 10.1097/YPG.0b013e3281ac2345. PMID 17728668
- [Background] Meltzer HY, Brennan MD, Woodward ND, Jayathilake K. Association of Sult4A1 SNPs with psychopathology and cognition in patients with schizophrenia or schizoaffective disorder. Schizophr Res. 2008 Dec;106(2-3):258-64. doi: 10.1016/j.schres.2008.08.029. Epub 2008 Sep 27. PMID 18823757
- [Background] Leucht S, Arbter D, Engel RR, Kissling W, Davis JM. How effective are second-generation antipsychotic drugs? A meta-analysis of placebo-controlled trials. Mol Psychiatry. 2009 Apr;14(4):429-47. doi: 10.1038/sj.mp.4002136. Epub 2008 Jan 8. PMID 18180760
- [Background] Wu EQ, Birnbaum HG, Shi L, Ball DE, Kessler RC, Moulis M, Aggarwal J. The economic burden of schizophrenia in the United States in 2002. J Clin Psychiatry. 2005 Sep;66(9):1122-9. doi: 10.4088/jcp.v66n0906. PMID 16187769
- [Background] Ascher-Svanum H, Zhu B, Faries D, Landbloom R, Swartz M, Swanson J. Time to discontinuation of atypical versus typical antipsychotics in the naturalistic treatment of schizophrenia. BMC Psychiatry. 2006 Feb 21;6:8. doi: 10.1186/1471-244X-6-8. PMID 16504026